CLINICAL TRIAL: NCT05721287
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of SBS-1000 Administered by Intravenous Infusion to Healthy Adult Subjects
Brief Title: A Phase 1, Randomized, Placebo-Controlled Safety and Tolerability Study Of Intravenous SBS-1000 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sparian Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBS1000-AP-101
Record Dates: First submitted 2023-01-31; First posted 2023-02-10 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pain; Acute Pain
Keywords: Arylepoxamide; Safety; Tolerability; SBS-1000; SBS1000; 6TM; AEAr Agonist
MeSH Terms: conditions — Pain; Acute Pain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SBS-1000 (Active Comparator): Investigational Product
  Interventions: Drug: SBS-1000
- Placebo (Placebo Comparator): Normal saline (0.9% sodium chloride [NaCl])
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SBS-1000 — SBS-1000 administered as a single continuous IV infusion over 60 minutes
  Other Names: arylepoxamide agonist
  Arms: SBS-1000
Drug: Placebo — Normal saline (0.9% sodium chloride [NaCl]) administered as a single dose IV infusion over 60 minutes
  Other Names: sodium chloride
  Arms: Placebo

SUMMARY:
This study will be a single-center, double-blind, randomized placebo-controlled, adaptive, single ascending dose study.

DETAILED DESCRIPTION:
This study will be a single-center (clinical research unit), double-blind, placebo-controlled, randomized, adaptive, single-ascending dose study receiving either Investigational Product (IP [SBS-1000]) or placebo IV infusion. Up to 56 subjects will be randomized.

A total of 6 ascending dose cohorts will be used to assess the MTD of SBS-1000. Each cohort will be comprised of up to 8 subjects randomized 6:2 (IP:placebo). A sentinel group of 2 subjects randomized 1:1 (IP:placebo) will be used for each cohort with the sentinel group being dosed at least 48 hours prior to dosing the remaining subjects of the cohort, and contingent on the results of ongoing safety evaluation.

Blood samples will be collected over 72 hours postdose and urine samples over 48 hours postdose for pharmacokinetic (PK) assessments in all cohorts. Pharmacodynamic assessments will be performed throughout the study in cohorts 1 through 6. The sampling parameters may be adjusted based on the interim safety review.

Once the maximum tolerated dose (MTD) is established, dosing with the MTD or a lower dose, as determined by an interim safety review, an additional cohort (7) will occur to investigate the cardiodynamic effects of SBS-1000 using Holter monitoring. Cohort 7 will be comprised of 8 subjects randomized 6:2 (IP:placebo). No sentinel dosing administration will occur in this cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Healthy adult male or female, aged 18 to 59 years, inclusive, at Screening
3. Body mass index (BMI) within 18.0 kg/m^2 to 33.0 kg/m^2, inclusively
4. Minimum body weight of at least 50.0 kg at Screening
5. Willingness to comply with all study procedures
6. If female, agrees to use an acceptable contraceptive method.
7. If male, agrees to use an acceptable contraceptive method.
8. Healthy as determined by no clinically significant findings at screening and clinic admission.
9. Non- or ex-smoker

Exclusion Criteria:

1. Has a current medical condition that would affect sensitivity to cold or pain
2. Personal or family history of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, dermatologic, or other clinically significant disease that may interfere with the study
3. Any clinically significant illness in the 28 days prior to the first study drug administration
4. Use of any prescription drugs in the 28 days prior to the first study drug administration, that in the opinion of an investigator would put into question the status of the participant as healthy
5. Routine or chronic use of acetaminophen and/or nonsteroidal anti-inflammatory drugs (NSAIDs)
6. Any clinically significant laboratory results at screening or prior to the first drug administration
7. intake of an investigational product within 28 days prior to study drug administration.
8. Positive test for alcohol and/or drugs of abuse
9. Positive for HIV or hepatitis
10. Donation of plasma 7 days prior to study drug administration and/or donation of blood within 56 days prior to study drug administration.
11. Significant ECG abnormalities

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | From start of infusion to 4 (±2) days after the last blood draw in the study
  Adverse events as assessed by electrocardiogram, vital signs, end-tidal carbon dioxide, oxygen saturation, physical examination, clinical laboratory tests, OAAS, C-SSRS, slit-lamp examination, gastrointestinal/esophageal assessment and concomitant medications

SECONDARY OUTCOMES:
Area under the plasma concentration (AUC) and Cmax versus time curve of SBS-1000 | From start of infusion to 72 hours post-infusion
  Assessment of systemic pharmacokinetics (PK) and urinary excretion of SBS-1000 by evaluation of AUC, Cmax, tmax, Ke t 1/2, Cl, V and Urine PK

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Reich, MD, Study Director — Sparian Biosciences
Locations (1):
- Altasciences Clinical Kansas, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No